CLINICAL TRIAL: NCT01503424
Title: An Open Label, Balanced, Randomized, Two-treatment, Two-period, Two-sequence, Single Oral Dose, Crossover, Bioequivalence Study of Olanzapine Tablets 5 mg With Zyprexa® Tablets 5 mg in Healthy Subjects Under Fed Conditions
Brief Title: Bioequivalence Study of Olanzapine Tablets, 5 mg Under Fed Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dr. Reddy's Laboratories Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 379-11
Record Dates: First submitted 2012-01-02; First posted 2012-01-04 (Estimated); Last update posted 2012-01-05 (Estimated); Status verified 2012-01

CONDITIONS: Fed
MeSH Terms: conditions — Lecithin Cholesterol Acyltransferase Deficiency | interventions — Olanzapine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Olanzapine Tablets, 5 mg (Experimental): Olanzapine Tablets, 5 mg of Dr. Reddy's Laboratories Limited
  Interventions: Drug: Olanzapine
- Zyprexa (Active Comparator): Zyprexa Tablets, 5 mg of Eli Lilly and company
  Interventions: Drug: Olanzapine

INTERVENTIONS:
Drug: Olanzapine — Olanzapine Tablets, 5 mg
  Other Names: Zyprexa

SUMMARY:
The purpose of this study is to compare the bioequivalence and characterize the profile of the olanzapine tablets, 5 mg with zyprexa tablets, 5 mg in healthy, adult, human subjects under fed conditions and to monitor the adverse events and ensure the safety of the subjects.

DETAILED DESCRIPTION:
An open label, balanced, randomized, two-treatment, two-period, two-sequence, single oral dose, crossover, bioequivalence study of Olanzapine Tablets 5 mg of Dr. Reddy's Laboratories Limited, India, comparing with that of Zyprexa® (Olanzapine) Tablets 5 mg of Eli Lilly and Company, USA, in healthy, adult, human subjects under fed conditions.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, adult, human volunteers between 18 and 45 years of age (both inclusive) living in and around Ahmedabad city of western part of IndIa.
* Having a Body Mass Index (BMI) between 18.5 and 24.9(both inclusive), calculated as weight in kg/height in m2.
* Non-smokers since at least six months.
* Have no significant diseases or clinically significant abnormal findings during screening,medical history, clinical examination, laboratory evaluations, 12- lead ECG and X-ray chest (postero-anterior view) recordings.
* Able to understand and comply with the study procedures. in the opinion of the Principal investigator.
* Able to give voluntary written informed consent for participation in the trial.
* In case of female subjects:

  * Surgically sterilized at least 6 months prior to study participation or
  * If of child bearing potential is willing to use a suitable and effective double barrier contraceptive method or intra uterine device during the study.
  * Pregnancy test must be negative.

Exclusion Criteria:

* Known hypersensitivity or idiosyncratic reaction to olanzapine to any of its excipients or any drug or any substance.
* History or presence of any disease or condition which might compromise the haemopoietic,renal, hepatic, endocrine, pulmonary, central nervous, cardiovascular, immunological, dermatological, gastrointestinal or any other body system.
* A recent history of harmful use of alcohol(less than 2 years),ie alcohol consumption of more than 14 standard drinks per week for men and 07 standard drinks per week for women (A standard drink is defined as 360 ml of beer or 150 ml of wine or 45 ml of 40% distilled spirits such as rum, whisky, brandy etc), or consumption of alcohol or alcoholic product within 48 hrs prior to receiving IMP.
* Inability to remain in an upright position at the time of dosing.
* Sitting blood pressure less than 110/70 mm Hg or pulse rate less than 60 or more than 100 beats per minute at the time of screening.
* Presence of orthostatic hypotension at the time of screening.
* Ingestion or Use of any medication at any time within l4 days prior to dosing in period-1. In any such case subject selection will be at the discretion of the Principal Investigator.
* Any history or presence of asthma (including aspirin induced asthma) or nasal polyp or NSAII)induced urticaria.
* Consumption of Grape fruits or its products within a period of 48 hours prior to receiving the study drug.
* The presence of clinically significant abnormal laboratory values during screening.
* Use of any recreational drugs or history of drug addiction or testing positive in pre-study drug scans.
* History or presence of psychiatric disorders.
* A history of difficulty with donating blood.
* Donation of blood (l unit or 350 mL) or receipt of an investigational medicinal product or participation in a drug research study within a period of 90 days prior to the first dose of study medication. Elimination half-life of the study drug should be taken into consideration for inclusion of the subject in the study.

Note: In case the blood loss is ≤ 200 mL; subject may be enrolled 60 days after blood donation or last sample of the previous study.

* A positive hepatitis screen including hepatitis B surface antigen and HCV antibodies.
* A positive test result for HIV antibody.
* An unusual diet, for whatever reason (e.g. low-sodium), for four weeks prior to receiving the study drug. In any such case subject selection will be at the discretion of the Principal Investigator.
* Nursing mothers (females).

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2011-08; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Bioequivalence is based on Cmax and AUC parameters | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Alpeshkumar Patel, MD, Principal Investigator — Lambda Therapeutic Research Ltd.
Locations (1):
- Lambda Therapeutic Research Ltd.,, Ahmedabad, Gujarat, India